CLINICAL TRIAL: NCT02937584
Title: A Randomized, Double-Blind, Two Treatment, Two Period, Chronic Dosing (2 Weeks), Cross-Over, Multi-Center Study to Evaluate the Effects of PT001 and PT005 on Specific Image Based Airway Volumes and Resistance in Subjects With Moderate to Severe COPD.
Brief Title: A Study to Assess the Effects of PT001 and PT005 MDI on Specific Image Based Parameters in Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT003019
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-06

CONDITIONS: COPD, Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GP MDI (PT001) 14.4 μg (Experimental): Glycopyrronium
  Interventions: Drug: GP MDI (PT001) 14.4 μg
- FF MDI (PT005) 9.6 μg (Experimental): Formoterol Fumarate
  Interventions: Drug: FF MDI (PT005) 9.6 μg

INTERVENTIONS:
Drug: GP MDI (PT001) 14.4 μg — Glycopyrronium
  Arms: GP MDI (PT001) 14.4 μg
Drug: FF MDI (PT005) 9.6 μg — Formoterol Fumarate
  Arms: FF MDI (PT005) 9.6 μg

SUMMARY:
To assess the effect of treatment with Glycopyronnium (GP) MDI administered twice daily (BID) and Formoterol Fumarate (FF) MDI administered BID on specific image-based airway volumes and resistance in subjects with moderate to severe chronic obstructive pulmonary disease (COPD) following chronic dosing after approximately two weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative urine pregnancy test at Visit 1, and agrees to use acceptable contraceptive methods used consistently and correctly
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* At Visit 1, FEV1/FVC ratio must be <0.70
* At Visit 1, post-bronchodilator FEV1must be >30% and <80% predicted normal value, calculated using The Third National Health and Nutrition Examination Survey (NHANES III) reference equations.

Exclusion criteria:

* Significant diseases other than COPD, i.e., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Visit 1 (Screening) or during the run-in period (Visit 1 to Visit 2).
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Visit 1 (Screening) or during the run-in period (Visit 1 to Visit 2).
* Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated.
* Subjects who have a history of hypersensitivity to β2-agonists, glycopyrronium or other muscarinic anticholinergics, or any component of the MDI.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Orevillo, Study Director — Pearl Therapeutics
Locations (2):
- Belgium (2):
  - Research Site, Edegem
  - Research Site, Erpent

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4186&filename=PT003019-01_FLUI-2015-140_Protocol_10%20August_Redacted_PDFA.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4186&filename=PT003019-sap-16APR2018-Redacted_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study randomized 23 subjects at 2 sites in Belgium from December 2016 to May 2018.
Pre-assignment Details: Subjects were randomized into 1 of 2 treatment sequences. Sequence 1 received GP MDI in Period 1 followed by FF MDI in Period 2. Sequence 2 received FF MDI in Period 1 followed by GP MDI in Period 2.
Groups:
- GP MDI/ FF MDI: Glycopyrronium Metered Dose Inhalation /Formoterol Fumarate Metered Dose Inhalation
- FF MDI/GP MDI: Formoterol Fumarate Metered Dose Inhalation / Glycopyrronium Metered Dose Inhalation
Period: Period 1
Arm/Group | GP MDI/ FF MDI | FF MDI/GP MDI
Started | 11 | 12
Completed | 10 | 10
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2
Period: Washout
Arm/Group | GP MDI/ FF MDI | FF MDI/GP MDI
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | GP MDI/ FF MDI | FF MDI/GP MDI
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population - all subjects who were randomized to treatment. Treatment was assigned as randomized regardless of the treatment actually received.
Groups:
- Overall Study: ITT Population
Arm/Group | Overall Study
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: ITT Population
  Years | 64.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Female | 6
    Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 23
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Specific Image-Based Airway Volume (siVaw)
Description: Specific image-based airway volume. Average across lobe, adjusted for lobe volume. Ratio to baseline
Time Frame: Baseline, Day 15
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- GP MDI: Glycopyrronium Metered Dose Inhalation
- FF MDI: FF MDI Formoterol Fumarate Metered Dose Inhalation
Arm/Group | GP MDI | FF MDI
Number analyzed (Participants) | 19 | 19
ratio | 1.11 [1.02 to 1.22] | 1.23 [1.14 to 1.33]
Statistical Analysis 1: Comparison: GP MDI; Test type: Other; p = 0.0187, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.11, 95% CI 2-sided [1.02 to 1.22]
Statistical Analysis 2: Comparison: FF MDI; Test type: Other; p < 0.0001, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.23, 95% CI 2-sided [1.14 to 1.33]

2. Primary Outcome: Specific Image-based Airway Resistance (siRaw)
Description: Specific image-based airway resistance (siRaw). Average across lobes, adjusted for lobe volume. Ratio to baseline.
Time Frame: Baseline, Day 15
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | GP MDI | FF MDI
Number analyzed (Participants) | 19 | 19
ratio | 0.75 [0.59 to 0.95] | 0.56 [0.44 to 0.71]
Statistical Analysis 1: Comparison: GP MDI; Test type: Other; p = 0.0219, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.75, 95% CI 2-sided [0.59 to 0.95]
Statistical Analysis 2: Comparison: FF MDI; Test type: Other; p < 0.0001, t-test, 2 sided — Statistical significance assessed using Hochberg's procedure applied across primary endpoints within each treatment; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.56, 95% CI 2-sided [0.44 to 0.71]

3. Secondary Outcome: Image-based Airway Volume (iVaw)
Description: Image-based airway volume (iVaw) without correction for lobe volume. Ratio to baseline.
Time Frame: Baseline, Day 15
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | GP MDI | FF MDI
Number analyzed (Participants) | 19 | 19
ratio | 1.12 [1.01 to 1.24] | 1.21 [1.12 to 1.31]
Statistical Analysis 1: Comparison: GP MDI; Test type: Other; p = 0.0283, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.12, 95% CI 2-sided [1.01 to 1.24]
Statistical Analysis 2: Comparison: FF MDI; Test type: Other; p < 0.0001, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 1.21, 95% CI 2-sided [1.12 to 1.31]

4. Secondary Outcome: Image-based Airway Resistance (iRaw)
Description: Image-based airway resistance (iRaw) without correction for lobe volume. Ratio to baseline.
Time Frame: Baseline, Day 15
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | GP MDI | FF MDI
Number analyzed (Participants) | 19 | 19
ratio | 0.76 [0.59 to 0.97] | 0.55 [0.41 to 0.72]
Statistical Analysis 1: Comparison: GP MDI; Test type: Other; p = 0.0304, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.76, 95% CI 2-sided [0.59 to 0.97]
Statistical Analysis 2: Comparison: FF MDI; Test type: Other; p = 0.0003, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.55, 95% CI 2-sided [0.41 to 0.72]

5. Secondary Outcome: FEV1
Description: FEV1 Change from baseline in Forced Expiratory Volume at 1 second.
Time Frame: Baseline, Day 15
Population: ITT Population
Measure: Mean (Standard Deviation); unit: L
Arm/Group | GP MDI | FF MDI
Number analyzed (Participants) | 19 | 19
L | 0.065 (0.193) | 0.151 (0.293)
Statistical Analysis 1: Comparison: GP MDI; Test type: Other; p = 0.1582, t-test, 2 sided; Within-group comparison to baseline using paired test; Mean Change from Baseline = 0.065, 95% CI 2-sided [-0.028 to 0.158]
Statistical Analysis 2: Comparison: FF MDI; Test type: Other; p = 0.0375, t-test, 2 sided; Within-group comparison to baseline using paired test; Mean Change from Baseline = 0.151, 95% CI 2-sided [0.010 to 0.292]

6. Secondary Outcome: Functional Residual Capacity (FRC)
Description: Functional residual capacity (FRC). Ratio to baseline.
Time Frame: Baseline, Day 15
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | GP MDI | FF MDI
Number analyzed (Participants) | 19 | 19
ratio | 0.978 [0.891 to 1.073] | 0.938 [0.833 to 1.056]
Statistical Analysis 1: Comparison: GP MDI; Test type: Other; p = 0.6176, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.978, 95% CI 2-sided [0.891 to 1.073]
Statistical Analysis 2: Comparison: FF MDI; Test type: Other; p = 0.2699, t-test, 2 sided; Within-group comparison to baseline using paired test; Geometric mean ratio to baseline = 0.938, 95% CI 2-sided [0.833 to 1.056]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent throughout the treatment period and up to 14 days following the last dose of study drug.
Description: The Safety Population was defined as all subjects who were randomized to treatment regardless and received at least one dose of study treatment. Serious adverse events collected from the time the subject signed consent up to 14 days following the last dose of study drug.
Arm/Group | GP MDI | FF MDI
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/22
Other Adverse Events (participants affected / at risk) | 3/20 | 3/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI (N=20) | FF MDI (N=22)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI (N=20) | FF MDI (N=22)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02937584/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT02937584/SAP_001.pdf